CLINICAL TRIAL: NCT00443079
Title: A Single-center, Single-blinded, Placebo-controlled Pilot Study of IdB 1016 (Siliphos) in Adult Patients With Non-alcoholic Steatohepatitis (NASH)
Brief Title: A Study of Siliphos in Adults With Non-alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heather Patton (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Sponsor-Investigator, Heather Patton, Professory, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 051117
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Fatty Liver
Keywords: Clinical Trials; Pilot Projects; Milk Thistle; Liver Function Tests
MeSH Terms: conditions — Fatty Liver | interventions — IdB 1016

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Siliphos/Placebo (Experimental): Received study medication first followed by placebo
  Interventions: Drug: IdB 1016 (Siliphos); Drug: Matched placebo
- Placebo/Siliphos (Experimental): Received placebo first followed by study medicaiton
  Interventions: Drug: IdB 1016 (Siliphos); Drug: Matched placebo

INTERVENTIONS:
Drug: IdB 1016 (Siliphos) — 1 pill 3 times daily x 6 weeks
Drug: Matched placebo — 1 pill 3 times daily x 6 weeks

SUMMARY:
The purpose of this study is to evaluate the dietary supplement Siliphos, which comes from milk thistle, to determine whether it is safe and well-tolerated in adults who have non-alcoholic steatohepatitis (NASH). An additional aim of this study is to determine whether Siliphos may be beneficial in treatment of NASH as indicated by improvement in liver enzymes (ALT and AST). The study hypothesis is that Siliphos will be safe and well-tolerated in people with NASH and will result in a decrease in the liver enzymes ALT and AST.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) encompasses a spectrum of liver conditions characterized by fat accumulation in the liver. Non-alcoholic steatohepatitis (NASH) is one form of NAFLD that may progress to cirrhosis in some people. Currently, there are no medications that are approved for the treatment of NASH. Milk thistle is sold over-the-counter as a dietary supplement. Milk thistle has been used for hundreds of years as a supplement to support liver function, and is commonly taken by people with a variety of liver conditions. Milk thistle may help to reduce inflammation and fibrosis (scar tissue) in the liver, so it may be beneficial in the treatment of NASH. As NAFLD is very common in the population, there are probably many people with NAFLD taking milk thistle supplements. However, there are no published studies of milk thistle in NAFLD. Therefore, this study is designed to provide preliminary evidence of the safety, tolerability, and efficacy of milk thistle in people with NASH.

Comparison: The milk thistle supplement (called Siliphos) will be compared to a placebo (sugar pill) in this study.

ELIGIBILITY:
Inclusion Criteria:

* Liver biopsy within 12 months demonstrating NASH
* Abnormal ALT

Exclusion Criteria:

* Uncontrolled diabetes
* Hepatitis B, hepatitis C, or other chronic liver conditions
* Abnormal kidney function
* Excess alcohol consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Patton, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego Medical Center, San Diego, California, United States

REFERENCES:
- [Background] Kidd P, Head K. A review of the bioavailability and clinical efficacy of milk thistle phytosome: a silybin-phosphatidylcholine complex (Siliphos). Altern Med Rev. 2005 Sep;10(3):193-203. PMID 16164374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with biopsy-proven NASH were recruited from outpatient hepatology clinics. Liver biopsy had to be within the previous year (no liver biopsies were done specifically to enroll in the study). ALT was elevated (normal ALT defined as 30U/L for men and 20U/L for women) and other types of chronic liver disease (viral hepatitis, alcohol, autoimmune) evaluated and excluded. Baseline kidney function was also normal (creatinine less than or equal to 1).
Pre-assignment Details: There were no participants who were excluded from study between informed consent/screening visit and study group allocation/randomization.
Groups:
- Siliphos/Placebo: Subjects treated with study drug (IdB 1016 1 pill by mouth 3 times daily) for 6 weeks with 2 weeks of washout followed by placebo 1 pill by mouth three times daily for 6 weeks
- Placebo/Siliphos: Subjects treated with placebo 1 pill by mouth three times daily for 6 weeks with 2 weeks of washout followed by study drug (IdB 1016 1 pill by mouth 3 times daily) for 6 weeks
Period: Overall Study
Arm/Group | Siliphos/Placebo | Placebo/Siliphos
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Siliphos/Placebo: Subjects treated with Siliphos (1 pill by mouth three times daily) for 6 weeks with 2 weeks of washout followed by placebo (1 pill by mouth three times daily) for 6 weeks
- Placebo/Siliphos: Subjects treated with Placebo (1 pill by mouth three times daily) for 6 weeks with 2 weeks of washout followed by Siliphos (1 pill by mouth three times daily) for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Siliphos/Placebo | Placebo/Siliphos | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Customized [Number; unit: participants]
  Age <50 years | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 3 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants With Adverse Events
Description: Side effect profile was collected at each study visit as tracked by study participants. Any new onset symptoms reported by study participants were recorded as side effects of treatment and analyzed according to whether they occurred while participants were treated with placebo or Siliphos.
  An increase in ALT value to greater than or equal to 2 x baseline value was also evaluated for possible drug induced liver injury.
Time Frame: 6 weeks
Population: side effects and adverse events were gathered from study participants at each clinic visit
Measure: Count of Participants; unit: Participants
Groups:
- Siliphos: All participants received both study drug and placebo. Adverse events were evaluated for all participants during the time period that they were receiving Siliphos.
  IdB 1016 (Siliphos): 1 pill 3 times daily x 6 weeks
- Placebo: Adverse events were evaluated for all participants during the time period that they received placebo.
  Placebo: 1 pill 3 times daily x 6 weeks
Arm/Group | Siliphos | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With a Decrease in ALT Value Greater Than or Equal to 15 U/L From Baseline to the End of the Treatment Era
Description: Change in ALT value from baseline to end of treatment arm during the time treated with Placebo in comparison to the time treated with Siliphos. Significant change in ALT was defined as a decrease by 15 or more units from baseline to end of treatment period.
Time Frame: 6 weeks
Population: Number participants with a decrease in ALT value greater than or equal to 15 U/L from baseline to the end of the treatment era.
Measure: Count of Participants; unit: Participants
Groups:
- Siliphos: Entire study population receiving 1 or more doses of study drug. Comparison of ALT measured at the beginning and end of treatment period during the time that Siliphos was administered.
  Siliphos 1 pill by mouth three times daily x 6 weeks
- Placebo: Entire study population receiving 1 or more doses of study drug. Comparison of ALT measured at the beginning and end of treatment period during the time that placebo was administered.
  Placebo 1 pill by mouth three times daily x 6 weeks
Arm/Group | Siliphos | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the beginning of the treatment through the end of follow-up (at time of last clinic visit, week 16 or 2 weeks after end of medication administration).
Description: Study participants were given journals to record any symptoms that may have emerged during treatment and asked to bring these with them to each study visit for investigator review and recording. Additional details about symptoms to be reviewed during study visits with investigator as they occur.
Groups:
- Siliphos: Siliphos 1 pill by mouth three times daily for 6 weeks (combined for all participants)
- Placebo: Placebo 1 pill by mouth three times daily for 6 weeks (combined for all participants)
Arm/Group | Siliphos | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No